CLINICAL TRIAL: NCT01418053
Title: Randomised Controlled Study on the Effect of a Kneipp Hot Cataplasm With Caraway Oil in the Treatment of Irritable Bowel Syndrome
Brief Title: The Effect of Hot Cataplasm With Caraway Oil in the Treatment of Irritable Bowel Syndrome
Acronym: CarO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-4627 CarO
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — caraway oil; Olive Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hot Cataplasm with Caraway Oil (Experimental)
  Interventions: Drug: caraway oil
- Hot Cataplasm with Olive oil (Active Comparator)
  Interventions: Drug: Olive oil
- Cold cataplasm with Olive oil (Active Comparator)
  Interventions: Drug: Olive oil

INTERVENTIONS:
Drug: caraway oil — essential oil, Carum carvi, 2% dissolved in olive oil, 1 teaspoon with caraway oil used externally as inunction together with a hot cataplasm
  Arms: Hot Cataplasm with Caraway Oil
Drug: Olive oil — 1 teaspoon with caraway oil used externally as inunction together with a hot or cold cataplasm as assigned
  Arms: Cold cataplasm with Olive oil; Hot Cataplasm with Olive oil

SUMMARY:
The purpose of this study is to determine whether a daily use of a Kneipp hot cataplasm with caraway oil is effective in the treatment of abdominal pain and complaints caused by Irritable bowel syndrome.

DETAILED DESCRIPTION:
see above.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome according to Rom-III
* Subtype Diarrhea or Alternating
* discomfort or pain > 1 times a week
* discomfort or pain > 4 on a Visual Analog Scale

Exclusion Criteria:

* Inflammatory bowel diseases (test results necessary)
* Lactose, Fructose Malabsorption (test results necessary)
* Celiac Disease
* Pregnancy or Breastfeeding
* Colectomy or Hemicolectomy >50cm
* Severe metabolic disorders, hormonal disorders, cardiac or respiratory failure, liver or renal diseases
* severe depression, psychotic or psychiatric disorders, substance abuse
* cancer within the last 5 years
* allergy to caraway
* acute inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome - Symptom Severity Score | at T2 (Day 21)
  IBS-SSS (Francis 1997)

SECONDARY OUTCOMES:
Frequency of abdominal discomfort/Pain | last week of treatment (days 14-21)
  Diary, daily rating of pain
Intensity of abdominal discomfort/Pain | last week of treatment (days 14-21)
  Daily rating of pain intensity on a 100mm Visual analogue scale, pain diary
Quality of life | T2 (Day 21)
  measured with the EQ-5D
Quality of life - ibs specific | T2 (day 21)
  measured with the IBS-QOL (Patrick, 1998)
Depression and Anxiety | T2 (day 21)
  HADS questionnaire (Hermann, 1995)
Global improvement | At day 7, 14 and 21
  Question on global improvement: How have your symptomes changed compared to the last week: from much worse to much better on a 7-point scale
h-BD2 | T2 (day 21)
  h-BD2 laboratory findings
Adequate Relief Score | at day 7, 14, 21
  Adequate Relief Score (Mangel, 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, MD, Prof, Principal Investigator — University Duisburg-Essen, Chair of Integrative Gastroenterology
Locations (1):
- Klinik für Naturheilkunde und Integrative Medizin, Essen, Germany

REFERENCES:
- [Result] Lauche R, Janzen A, Ludtke R, Cramer H, Dobos G, Langhorst J. Efficacy of Caraway Oil Poultices in Treating Irritable Bowel Syndrome--A Randomized Controlled Cross-Over Trial. Digestion. 2015;92(1):22-31. doi: 10.1159/000398790. Epub 2015 Jun 5. PMID 26044145